CLINICAL TRIAL: NCT06754618
Title: The Influences of Single Chamber Vs. Multi-chamber Blood Flow Restriction Biceps Curls on Acute Arterial Stiffness, Perceptual Responses and Performance
Brief Title: The Influences of Single Chamber Vs. Multi-chamber Blood Flow Restriction Cuffs with Bicep Curls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salisbury University (Other)
Responsible Party: Principal Investigator, Timothy Werner, Professor, Salisbury University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 364
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Blood Vessel Disease; Muscle Edema
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will undergo three treatment sessions (no BFR, SC BFR, and MC BFR) in a randomized order separated by one week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- single chamber blood flow restriction cuff (Experimental): Single Chamber BFR (Delfi, Vancouver, Canada) training devices will be used for exercise and testing sessions (see attachment). Cuffs will be placed around the right and left proximal arm. The LOP will be set at 60% immediately before exercise and will be applied during the entire exercise set (approximately 30-60 seconds in duration) in accordance with manufacturer specifications. The cuffs will maintain pressure during training and rest periods. The LOP will be decreased to 0% immediately after the set is completed.
  Interventions: Device: Delfi
- Multiple chamber blood flow restriction cuff (Experimental): Multiple chamber BFR (B-Strong, Park City, UT) training devices will be used for exercise and testing sessions (see attachment). Cuffs will be placed around the right and left proximal arm. The LOP will be set at 60% immediately before exercise and will be applied during the entire exercise set (approximately 30-60 seconds in duration) in accordance with manufacturer specifications. The cuffs will maintain pressure during training and rest periods. The LOP will be decreased to 0% immediately after the set is completed.
  Interventions: Device: Delfi
- No BFR cuff (Placebo Comparator): No cuff will be worn during the training session.
  Interventions: Device: Delfi

INTERVENTIONS:
Device: Delfi — Cuffs will be worn throughout the entire training session. Training session consist of lower intensity bicep curls. Four sets of wall squats will be performed to failure. Arterial stiffness and muscle morphological assessments will be conducted before and after the exercise.

SUMMARY:
The purpose of this study is to investigate the use of single (SC) and multi-chamber (MC) blood flow restriction (BFR) cuff bicep exercise on indices of arterial stiffness, muscle morphology, and participant perception.

DETAILED DESCRIPTION:
Twenty six adults aged 18-40 years old will undergo three treatment sessions (control (no BFR), SC BFR, and MC BFR) in a randomized order separated by one week. A familiarization session will also occur one week before starting the treatment period. Each subject will undergo a series of tests including anthropometry, ultrasonography of the carotid artery, applanation tonometry, ultrasonography of the vastus lateralis, blood pressure acquisition, body composition, and maximal strength assessments (1RM). The exercise trial will consist of sets of dumbbell bicep curls performed to failure with a 2-seconds concentric and 2-seconds eccentric cadence, at 20% of their 1RM using 60% of the supine limb occlusion pressure (LOP) with 1-minute rest intervals. Assessments will be performed immediately before and after the exercise bout during each treatment session. Two-way ANOVAs will be used to examine the main effects of treatment and treatment-order interaction on pulse wave velocity, muscle cross-sectional area, and perceptual response.

ELIGIBILITY:
Inclusion Criteria:

1. Physically active (> 1,000 MET/min/wk) for at least six months.
2. Weight stable for previous 6 months (+/-2.5 kg)
3. Female subjects only- reported regular menstrual cycles for the last 2 years

Exclusion Criteria:

1. BP>140/90 mmHg
2. BMI>40 kg/m2
3. Diabetes
4. Familial hypercholesterolemia
5. Past or current history of CHD, stroke or major CVD events. Respiratory diseases (not including asthma), endocrine or metabolic, neurological, or hematological disorders that would compromise the study or the health of the subject.
6. Women must not be pregnant, plan to become pregnant during the study, or be nursing
7. Active renal or liver disease
8. All medications and supplements that influence dependent variables*
9. Recent surgery < 2 months
10. Alcohol abuse
11. Sleep apnea
12. Claustrophobia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | Prior to and 10-minutes after the exercise intervention
  A measurement of vascular health.

SECONDARY OUTCOMES:
Muscle Morphology | Prior to and immediately after the exercise intervention
  A measurement of bicep brachii cross sectional area

CONTACTS AND LOCATIONS:
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data when requested.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared after study is published for five years.